CLINICAL TRIAL: NCT00126282
Title: A Randomized, Double-blind, Placebo-controlled Medication Trial With D-Cycloserine for Individuals With Obsessive-compulsive Disorder Currently Receiving Behavior Therapy
Brief Title: A Medication Trial Combined With Behavior Therapy for Individuals With Obsessive-compulsive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Sabine Wilhelm, Ph.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-P-0001325
Record Dates: First submitted 2005-08-02; First posted 2005-08-03 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2008-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; behavior therapy; D-Cycloserine; medication; treatment trial; placebo-controlled; double-blind; randomized
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Behavior Therapy; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: behavior therapy
Drug: D-Cycloserine

SUMMARY:
This study examines the efficacy of the medication D-Cycloserine in the reduction of obsessions and compulsions in individuals with obsessive-compulsive disorder (OCD). All study participants will receive Exposure and Response Prevention, a common form of behavior therapy for individuals with OCD. Half (50%) of the participants will be randomly assigned to the placebo condition and the other half (50%) will be randomly assigned to receive D-Cycloserine. Because all participants will receive 10 sessions of behavior therapy, all participants are expected to improve from this treatment.

DETAILED DESCRIPTION:
The study consists of Behavior Therapy (Exposure and Response Prevention; ERP) for OCD. Specifically, it involves exposure to anxiety-provoking situations and response-prevention of any rituals. ERP has shown to be effective for many individuals with OCD.

All assessments and treatment sessions are at no cost to the patients. 50% of the patients will randomly be assigned to the D-Cycloserine (DCS) condition, and 50% of the patients will be assigned to a placebo condition. D-Cycloserine is FDA-approved for the treatment of Tuberculosis. However, recent research in other anxiety disorders has shown that D-Cycloserine plus Behavior Therapy is more effective than Behavior Therapy alone.

This treatment study has two active conditions. That is, all patients will receive Behavior Therapy and we do expect that everybody will improve from this treatment. However, it may be that those patients in the DCS condition will improve somewhat more than those in the placebo condition.

The treatment will be structured with homework and repeated assessments every 4 weeks. Assessments are extremely important as they guide the treatment and provide the study investigators necessary information about the treatment. The treatment consists of 10 sessions (twice a week) plus post-treatment and follow-up assessments at 1 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnosis for obsessive-compulsive disorder

Exclusion Criteria:

* History of psychotic disorders
* History of neurological disorders
* History of bipolar disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-12; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
significant reduction of OCD symptoms after the completion of treatment

SECONDARY OUTCOMES:
significant reduction of depressive symptoms after the completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital; David Tolin, PhD, Principal Investigator — Hartford Institute of Living
Locations (2):
- United States (2):
  - Anxiety Disorders Center, The Institute of Living, Hartford, Connecticut
  - Massachusetts General Hospital, Boston, Massachusetts